CLINICAL TRIAL: NCT02722564
Title: Accuracy of Self-estimation of Blood Alcohol Concentration Compared to Object Values
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's Hospital and Health Network, Pennsylvania (Other)
Responsible Party: Principal Investigator, Holly Stankewicz, D.O., attending physician and faculty emergency medicine resiency, St. Luke's Hospital and Health Network, Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: SLHN 2015-26
Record Dates: First submitted 2015-10-16; First posted 2016-03-30 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Alcohol Intoxication
MeSH Terms: conditions — Alcoholic Intoxication | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- all study participants (Experimental): subject will self estimate breath alcohol content and their actual BrAC will be recorded as measured by the Alco Sensor IV after each beer ingested.
  Interventions: Behavioral: self estimation of breath alcohol content; Device: breath alcohol content as measured by Alco Sensor IV device; Other: drink a beer

INTERVENTIONS:
Behavioral: self estimation of breath alcohol content
Device: breath alcohol content as measured by Alco Sensor IV device
Other: drink a beer — drink a beer, repeat until breath alcohol content 0.1

SUMMARY:
This will be a prospective survey study. The participants will all be volunteers of legal drinking age. Each participant will consume one alcoholic beverage (beer) at a time and then will be asked to verbally estimate their current blood alcohol concentration and if the subject feels they are able to drive. At that time, their BAC level will be measured objectively using a breath alcohol test (BAT) device. The participant will not be told their objective value. This will continue with a verbal estimate and actual BAT reading after every drink until the participant reaches a minimum BAC of 0.10. At this time, participants will continue to be monitored until their BAC falls to 0.08 and they are clinically sober. As their blood alcohol level decreases, the investigators will ask the participant to estimate their level every hour along with an actual reading until reaching 0.08. Statistical analyses will be used to determine how accurate self estimation is in regards to blood alcohol content.

ELIGIBILITY:
Inclusion Criteria:

* over the legal age (21years old) to drink alcohol.

Exclusion Criteria:

* Volunteers will be excluded from the study if they suffer from any of the following conditions:

Alcoholism, Diabetes, Kidney/bladder stones, Kidney disease, Liver disease, Stomach ulcer, Organ transplant patients, Dialysis patients, and patients with alcohol allergies.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- St. Luke's University Hospital, Bethlehem, Pennsylvania, United States

REFERENCES:
- [Background] Kraus CL, Salazar NC, Mitchell JR, Florin WD, Guenther B, Brady D, Swartzwelder SH, White AM. Inconsistencies between actual and estimated blood alcohol concentrations in a field study of college students: do students really know how much they drink? Alcohol Clin Exp Res. 2005 Sep;29(9):1672-6. doi: 10.1097/01.alc.0000179205.24180.4a. PMID 16205367

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: subject will self estimate breath alcohol content after each beer ingested
  self estimation of breath alcohol content
  record breath alcohol content as measured by breathalyzer
  drink a beer: drink a beer, repeat until breath alcohol content 0.1
Period: Overall Study
Arm/Group | All Study Participants
Started | 55
Completed | 55
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 55
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Change in Breath Alcohol Content Between the Estimated Level and the Actual Level as Measured by an Alco Sensor IV Device
Description: The change was measured both when participants' breath alcohol content was ascending to 0.1 and descending to 0.08.
Time Frame: 1 day
Population: The number analyzed for ascending BrAC readings and descending BrAC readings
Measure: Median (Standard Deviation); unit: percent blood alcohol content
Units Other Than Participants: BrAC readings
Arm/Group | All Study Participants
Number analyzed (Participants) | 55
Number analyzed (BrAC readings) | 587
percent blood alcohol content
  BrAC ascending to 0.1: number analyzed (BrAC readings) | 354
  BrAC ascending to 0.1 | 0.01 (0.02)
  BrAC descending to 0.08: number analyzed (BrAC readings) | 233
  BrAC descending to 0.08 | -0.01 (0.04)
Statistical Analysis 1: Comparison: All Study Participants; Test type: Other; p < 0.001, t-test, 2 sided — p value associated with the change between estimated and actual BrAC when the participants BrAC was ascending to 0.1
Statistical Analysis 2: Comparison: All Study Participants; Test type: Other; p < 0.0001, t-test, 2 sided — p value associated with change between estimated and actual BrAC as participants BrAC descended to 0.08

ADVERSE EVENTS:
Time Frame: 12 hours
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 8/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=55)
vomiting (Gastrointestinal disorders) | 5 (5)
vertigo (Ear and labyrinth disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes